CLINICAL TRIAL: NCT05846750
Title: A Prospective, Open-label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of Obinutuzumab(GA101) in Combination With Lenalidomide in Relapsed and Refractory(R/R) Marginal Zone Lymphoma (MZL)
Brief Title: Obinutuzumab in Combination With Lenalidomide in Relapsed or Refractory Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDHMZL2023
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-03

CONDITIONS: Marginal Zone Lymphoma
Keywords: Obinutuzumab; Lenalidomide
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab and lenalidomide (Experimental): Patients will be treated with obinutuzumab and lenalidomide for 6 cycles as induction, and the patients who achieve at least a partial response after 6 cycles of induction therapy will be eligible to enter the maintenance phase for 2 years
  Interventions: Drug: Obinutuzumab; Drug: lenalidomide

INTERVENTIONS:
Drug: Obinutuzumab — Induction (6 cycles, every 28 days/cycle): 1000 mg each time, administered on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-6 ( 8 total infusions)；
  Maintenance(12 cycles, every 2 months/cycle): 12 infusions of 1000 mg every 2 months for 2 years or until disease progression
  Other Names: GA101
Drug: lenalidomide — Induction( 6 cycles, every 28 days/cycle): 20 mg/day, oral, Dosing on Days 2-22, every 28 days/cycle of Cycles 1-6；
  Maintenance(12 cycles, every 28 days/cycle):10 mg on Days 2-22 of each 28-day cycle, 12 cycles for 1 year or until disease progression

SUMMARY:
This is a prospective, multicenter clinical study that will enroll 59 patients with relapsed and refractory (R/R) MZL. The study is designed to evaluate the efficacy and safety of the combination of obinutuzumab and lenalidomide in the treatment of relapsed and refractory marginal zone lymphoma (MZL).

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is incurable, and the vast majority of patients with MZL eventually face disease relapse or progression.

There is no standard second-line treatment for relapsed/refractory MZL, and the synergistic effect of obinutuzumab and lenalidomide has been demonstrated in other indolent lymphomas.

The aim of this trial is to investigate the efficacy and safety of the combination of obinutuzumab (GA101) and lenalidomide in the treatment of R/R marginal zone lymphoma in order to find a safe and effective option for this type of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
4. Histologically confirmed MZL. have a definite diagnosis of MZL
5. Prior treatment with at least one line of systemic lymphoma including prior immunotherapy or chemoimmunotherapy
6. At least one bi-dimensionally measurable nodal lesion (> 1.5 cm in greatest diameter on CT scan or MRI) OR at least one bi-dimensionally measurable extranodal lesion (> 1.0 cm in greatest diameter on CT scan or MRI)
7. Need for systemic therapy as assessed by the investigator
8. Life expectancy ≥ 3 months
9. Adequate blood function (except for abnormalities considered by the investigator to be due to the underlying disease of lymphoma), defined as follows:

   Hemoglobin ≥ 7 g/dL; Absolute neutrophil count ≥ 1.0 × 109/L; Platelet count ≥ 50 x 109/L
10. Normal laboratory values:

    Creatinine clearance ≥ 30 mL/min; Glutathione transaminase(AST) or glutathione aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN); Serum bilirubin ≤ 2 × ULN (≤ 3 × ULN in patients with Gilbert's syndrome)
11. For men who are not surgically sterile: Agree to use barrier contraception during treatment and for at least 3 months after the last dose of obinutuzumab or lenalidomide or as required by institutional guidelines, whichever is longer. In addition, male patients must agree to have their partner use an alternative method of contraception (e.g., oral contraceptive, intrauterine device, barrier method, or spermicide)
12. For women who are not surgically sterile: use two appropriate methods of contraception, such as oral contraceptives, intrauterine device, or barrier methods, in combination with spermicide for at least 28 days prior to agreeing to start of study medication, during treatment and for at least 12 months after the last dose of either obinutuzumab or lenalidomide, or as required by institutional guidelines, whichever is longer -

Exclusion Criteria:

1. Patients who are refractory or resistant to lenalidomide or obinutuzumab, refractory is defined as no response (PR or CR) after the start of treatment, or relapse within 6 months (≤ 2 cycles of prior lenalidomide or obinutuzumab and no exclusion of treatment change for non-refractory reasons)
2. History of serious allergic or anaphylactic reactions to monoclonal antibody therapy
3. Known hypersensitivity to any of the study drugs
4. Known sensitivity to murine products
5. Previous ≥ Grade 3 allergic reactions/Hypersensitivity to thalidomide
6. History of erythema multiforme, Grade 3 rash, or blisters following prior immunomodulatory derivative therapy
7. Histologically transformed, highly malignant or diffuse large B-cell lymphoma
8. Central nervous system or meningeal involvement by lymphoma
9. Contraindications for the investigational medical product included in the study treatment regimen
10. Positive test for chronic hepatitis B infection (defined as positive HBsAg serology)
11. Hepatitis C positive (hepatitis C virus antibody serology)
12. HIV or Human T-Lymphocytic Leukemia Virus 1 (HTLV1) positive
13. Evidence of any serious, uncontrolled co-morbidities that affect compliance with the protocol or interpretation of results, including but not limited to significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmias, or unstable angina), or significant pulmonary disease (including history of obstructive pulmonary disease or bronchospasm)
14. Infection caused by known active bacteria, viruses, fungi, or other microorganisms (other than fungal infection of the nail bed), or any major infection requiring intravenous antibiotics or hospitalization (completion of the entire course of antibiotics, except for neoplastic fever) within 4 weeks prior to enrollment
15. Prior malignancy other than lymphoma, unless the subject has a disease-free survival of ≥ 5 years
16. Pregnant or lactating women.
17. Have ≥ Grade 2 neuropathy
18. Participation in another clinical trial using a pharmacological intervention during the trial or within 28 days prior to Cycle 1
19. Corticosteroids within 4 weeks of enrollment, unless administered at a dose equivalent to ≤ 30 mg/day prednisone (within 4 weeks)
20. Past history of progressive multifocal leukoencephalopathy (PML)
21. Live vaccines within 28 days of treatment start
22. History of solid organ transplantation
23. Presence of any serious illness or abnormality in the clinical laboratory test results that, in the opinion of the investigator, would make the patient unable to safely participate and complete this study, or affect protocol compliance or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate(ORR) | 24 weeks
  Disease response evaluation after 6 cycles will be used to determine the overall remission rate

SECONDARY OUTCOMES:
2-year Progression Free Survival (PFS24): | up to 4.5 years
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
2-year Event-Free Survival (EFS24) | up to 4.5 years
  Event-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse, initiation of new anti-lymphoma therapy or death from any cause.
Complete Response Rate (CR) | 24 weeks
  Disease response evaluation after 6 cycles will be used to determine the overall remission rate
Overall survival (OS) | up to 4.5 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause.
  Alive patients will be censored at their last date known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Dr, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tian, China

IPD SHARING:
Plan to Share IPD: No